CLINICAL TRIAL: NCT07223333
Title: First-in-Human, Randomized, Double-Blind, Placebo-Controlled Study of Single Ascending Doses in Healthy Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics of PATAS
Brief Title: A Study of PATAS Trifluoroacetate Using Single Ascending Doses in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AdipoPharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PATAS-CL-001
Record Dates: First submitted 2025-10-28; First posted 2025-10-31 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy subjects, Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Healthy Subjects, Active (Experimental)
  Interventions: Drug: PATAS Trifluoroacetate

INTERVENTIONS:
Drug: PATAS Trifluoroacetate — A drug targeting the interaction between the ALMS1 protein and alpha-PKC
  Arms: Healthy Subjects, Active
Drug: Placebo — Excipient only formulation, without active compound
  Arms: Healthy subjects, Placebo

SUMMARY:
The primary objective of this study is to evaluate safety and tolerability of single subcutaneous (SC) doses of PATAS in healthy subjects. The secondary objective of this study is to determine the pharmacokinetics (PK) of single SC doses of PATAS in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Single Ascending Dose Inclusion criteria

  1. Healthy male and female subjects, 18 to 55 years of age, inclusive, at the time of signing the Informed Consent Form (ICF);
  2. Willing and able to give written informed consent for participation in the study prior to the initiation of any Screening or study-specific procedures;
  3. Body mass index (BMI) within the range of 20.0 to 35.0 kg/m2, inclusive, at Screening;
  4. In generally good health, as judged by the Investigator, based upon medical/surgical history and the results of physical examination, vital signs, clinical laboratory assessments, and 12-lead electrocardiogram (ECG) at Screening and at Check-In (Day -1);
  5. Female subjects must have a negative serum pregnancy test result at the Screening Visit and a negative urine pregnancy test at Check-In (Day -1) (prior to the first dose of study drug) and must not be pregnant, lactating, or planning a pregnancy from the Screening Visit to 90 days after the last dose of study drug;
  6. Negative test result for severe acute respiratory syndrome coronavirus 2 at Check-In (Day -1); and
  7. Willing to comply with all study procedures and requirements throughout the duration of the study.

Exclusion Criteria:

1. Clinically significant history of asthma, eczema, or any other allergic condition or previous severe hypersensitivity; Note: Non-active hay fever is not exclusionary.
2. Liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase [ALP], total bilirubin) outside the following upper limits of normal (ULNs) at Screening or at Check-In (Day -1): a. For ALT and AST, measurements >1.5 × ULN; b. For ALP, measurements >2 × ULN; or c. For total bilirubin, measurements >1.5 × ULN.
3. Estimated glomerular filtration rate £60 mL/min/1.73 m2 based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at Screening or at Check-In (Day -1);
4. Thyroid-stimulating hormone (TSH) outside of reference range (e.g., TSH <1 × lower limit of normal [LLN] or TSH >1 × ULN) at Screening; Note: Abnormal TSH results will reflex to a free thyroxine (T4) test.
5. History of unexplained syncope, cardiac arrest, unexplained cardiac arrythmias or torsades de pointes, or structural heart disease;
6. Personal or family history of long QT syndrome;
7. Clinically significant history of any disease or disorder (i.e., gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric, or metabolic) deemed to be exclusionary, as judged by the Investigator;
8. Abnormal pulse rate or blood pressure (BP) measurements at Screening, defined as: a. Pulse rate <40 bpm or >100 bpm; b. Systolic BP <90 mmHg or >140 mmHg; or c. Diastolic BP <50 mmHg or >90 mmHg.
9. Clinically significant ECG abnormalities at Screening or at Check-In (Day -1), defined as prolongation of the average QTcF interval >450 ms for males and >470 ms for females, or other clinically significant ECG abnormalities per Investigator discretion;
10. Positive for hepatitis B surface antigen, HIV antibody, or hepatitis C virus antibody at Screening;
11. Receipt of any investigational product within 30 days prior to first study drug administration (90 days for investigational biologic agents) or 5 half-lives prior to first study drug administration, whichever is greater, or participation in >3 clinical studies within 12 months; 22. Known or suspected hypersensitivity to PATAS or any components of the formulation used (sodium hydroxide or mannitol);

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety -- 1A | 29 days
  Incidence and severity (using CTCAE version 5.0.) of treatment-emergent AEs and SAEs and evaluation of pharmacokinetic data

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Marion, Ph.D., Study Chair — AdipoPharma LLC
Locations (2):
- United States (2):
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio
  - Medpace Clinical Pharmaology Unit, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
This data is confidential.